CLINICAL TRIAL: NCT03094572
Title: Evaluation of the Visual Motor Task's Impact on the Behavior of a Neuronal and Spinal Network in Hemiplegic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2016-A01190-51
Record Dates: First submitted 2017-03-23; First posted 2017-03-29 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Human Spinal Cord Circuitry
Keywords: spinal cord circuitry; hemiplegia; rhythmic task
MeSH Terms: conditions — Hemiplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- visual motor tasks with dominant arm (1) (No Intervention): experimental arm for the first sub-study healthy volunteer
- control tasks with dominant arm (No Intervention): control arm for the first sub-study healthy volunteer
- visual motor tasks with non-dominant arm (No Intervention): control arm for the second sub-study healthy volunteer
- visual motor tasks on dominant arm, flexion movement (No Intervention): experimental arm for the third sub-study healthy volunteer
- visual motor tasks on dominant arm, extension movement (No Intervention): experimental arm for the third sub-study healthy volunteer
- visual motor tasks (Experimental): fourth sub-study with hemiplegic patient
  Interventions: Other: visual motor tasks
- visual motor tasks with dominant arm (2) (No Intervention): experimental arm for the second sub-study healthy volunteer

INTERVENTIONS:
Other: visual motor tasks — This exercise involves manipulating an object that corresponds to a "racket", this racket has a virtual avatar that animated a virtual ball. The purpose is to make it bounce to a given height. This comes close to ping-pong game.
  Arms: visual motor tasks

SUMMARY:
The general objective being to determine the modifications nature induced by upper extremity kinematic rhythmic task realization on cervical HSCC.

The obtained knowledge could open up new prospects for rehabilitation in cerebro-injured subjects in addition to existing therapeutics.

DETAILED DESCRIPTION:
Half of all stroke patients have physical disabilities. These disabilities combine sensory and motor deficiencies (control deficit, syncinesia, tone disorders) that cause disruption of upper extremity (UE) function (orientation, UE length adjustment and grip). The human spinal cord circuitry (HSCC) participate in the motion regulation. Roche et al. studied in healthy subjects the HSCC modifications during the visuo-motor regulation of the object clamping force by the hand. The authors showed that the learning of the task in a single session was associated with HSCC modifications, specific or not depending on the HSCC and according to a visual biofeedback associated or not to the task. Diserens et al. showed also that a rhythmic movement of UE pedaling causes a decrease in spasticity in hemiplegic subjects. Moreover, HSCC modification is dependent on the task performed. The rhythmic ball-bouncing in a virtual environment is a visuo-motor task rhythmic kinematic already studied in the healthy subject. To our knowledge, the present study is the first to investigate HSCC modification in hemiplegic subjects performing a rhythmic kinematic task with UE. We hypothesize that such a task leads to HSCC excitability specific modifications in the cervical spinal cord and leads to an improvement in the motor capabilities of the subjects.

The general objective being to determine the modifications nature induced by UE kinematic rhythmic task realization on cervical HSCC, our research will be broken down into four studies.

Study 1 will identify the influence of visual feedback on changes in HSCC excitability in a voluntary group. In this first study, 16 voluntary subjects will perform the visuo-motor task with their dominant UE and the control task (without visual feedback) with their dominant UE.

Study 2 will investigate the impact of UE laterality which performing the task on changes in HSCC excitability in a voluntary group. In this second study, 16 volunteer subjects will perform the visuo-motor task with their dominant UE and the visuo-motor task with their non-dominant UE.

Study 3 will objectify the effect of the type of contraction of the muscles involved in the task on changes in HSCC excitability in a volunteer group. In this third study, 16 voluntary subjects will perform the visuo-motor task with their dominant UE by performing either elbow flexion-extension or only flexion-extension of the wrist.

Finally, study 4 will study the effect of the pathology and the motor strategies used on the changes in HSCC excitability. In the latter study, 16 hemiplegic patients will perform the visuo-motor task with their paretic UE and spontaneous motor strategies.

The obtained knowledge could open up new prospects for rehabilitation in cerebro-injured subjects in addition to existing therapeutics.

ELIGIBILITY:
Inclusion Criteria:

Hemiplegic subjects:

* Informed consent signature,
* Male or female aged 18 years or over,
* Hemiplegic patient with single stroke,
* Patient able to stand without technical assistance,
* Patient capable of performing an active elbow flexion/extension movement of an amplitude of at least 45° against gravity,
* Patient able to understand and realize the cyclical kinematic rhythmic task.
* Absence of cognitive impairment, Mini-Mental State score (MMS) equal to 30.

Voluntary subjects:

* Informed consent signature,
* Male or female aged 18 years or over,

Exclusion Criteria:

Hemiplegic subjects:

* Refusal to participate in the study,
* Inability to cooperate,
* Intervention on the studied upper limb dating less than 6 months,
* No affiliation to a social security scheme,
* No H-reflex in the muscle Flexor Carpi Radialis,
* Epilepsy antecedent.in the year prior to inclusion.

Voluntary subjects:

* Refusal to participate in the study,
* Inability to cooperate,
* Intervention on the studied upper limb dating less than 6 months,
* No affiliation to a social security scheme,
* No H-reflex in the Flexor Carpi Radialis muscle,
* Ambidextrous subject,
* Epilepsy antecedent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2017-07-13 (Actual); Primary Completion 2018-07-23 (Actual); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Hoffmann's reflex amplitude | 2h
  amplitude modification of the hoffmann's reflex

SECONDARY OUTCOMES:
bell's test | 15 min
  The Bells Test is a cancellation test that allows for a quantitative and qualitative assessment of visual neglect
kinematic performance of the rhythmic task | 20 min
  task performance, learning task
modified Ashworth scale | 15 min
  spasticity evaluation
fugl meyer test | 40 min
  is an index to assess the sensorimotor impairment in individuals who have had stroke
MRC testing | 30 min
  muscle strengh mesurement

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas ROCHE, MD PhD, Principal Investigator — Raymond Poincare HOSPITAL
Locations (1):
- Nicolas ROCHE, Md PhD, Garches, France

IPD SHARING:
Plan to Share IPD: No